CLINICAL TRIAL: NCT01914042
Title: Prediction of Inter-individual Differences in the Response to Morphine by Psychophysical Assessment of Pain Enhancing and Inhibiting Mechanisms in Patients With Chronic Neuropathic Pain
Brief Title: Prediction of Inter-individual Differences in the Response to Morphine Versus Milnacipran in Patients With Sciatica
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Eisenberg Elon MD, Director, Pain Research Unit, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 143-10 RMB
Record Dates: First submitted 2013-07-22; First posted 2013-08-01 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Neuropathic Pain
Keywords: Opioid induced hyperalgesia; Neuropathic pain; Opioids; Sciatica; Serotonin-norepinephrine reuptake inhibitor (SNRI)
MeSH Terms: conditions — Neuralgia; Sciatica | interventions — Morphine; Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Experimental): Morphine in changing dosages (range between 10-60 mg twice a day). Opioid titration proceeds as follows: starting at an oral dose of 10 mg twice per day, followed every 5 days by a dose increase of 10 mg twice per day until (1) adequate analgesia had been achieved (as determined by the patients), (2) side effects (severe sedation, nausea or vomiting, constipation, sleep disturbances) limited further titration, or (3) a total of 120 mg per day had been reached.
  Interventions: Drug: Morphine
- Milnacipran (Active Comparator): Milnacipran (Ixel)- a serotonin-norepinephrine reuptake inhibitor (SNRI), will be administrated in changing dosages (range between 12.5-75 mg twice daily). SNRI titration proceeds as follows: starting at an oral dose of 12.5 mg twice per day, followed every 5 days by a dose increase of 12.5 mg twice per day until (1) adequate analgesia had been achieved (as determined by the patients), (2) side effects (severe sedation, nausea or vomiting, constipation, sleep disturbances) limited further titration, or (3) a total of 150 mg per day had been reached.
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Morphine
  Arms: Morphine
Drug: Milnacipran
  Arms: Milnacipran

SUMMARY:
Clinical, psychophysical, behavioral or genetic factor will predict the response to opioid treatment in patients with chronic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe chronic neuropathic pain or patients with radiculitis between 18 and 75 years of age.
2. Candidates for chronic opioid therapy for nonmalignant pain as determined by treating physician.
3. Patients treated with non-opioid analgetics, anti- inflammatory drugs or low opioid dosage (< 30 mg of oral morphine-equivalents per day).
4. Ability to understand the purpose and instructions of the study and to sign an informed consent.

   -

   Exclusion Criteria:

1.Diabetic Neuropathy 2.Pain in upper limbs 3.Receiving anti- depressants and/or anticonvulsants 4.Pregnant women 5.Inability to comply with study protocol. 6.Allergy to Opioids 7.A diagnosis of Raynaud's Syndrome 8.History of substance abuse

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain intensity (NPS) | 1 month

SECONDARY OUTCOMES:
Heat pain intensity in a remote area (Opioid induced hyperalgesia) | 1 month
  Heat pain sensitivity will be determined by the use of VAS units (0-100). We'll measure the intensity of pain in response to application of brief experimental heat pain.
The McGill Pain Questionnaire | At baseline and at the end of 4-week treatment period
  Will be completed before and after treatment
Assessment of Adverse events | Ongoing throughout the entire study period, an expected average of 4 weeks.
  A list of possible side effects from the administered drugs has been prepared and will be completed at all scheduled visits.
  In addition, patients will record AEs on daily basis. If needed patients can call and report adverse events by phone.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel